CLINICAL TRIAL: NCT05137197
Title: A Prospective, Randomized, Double-Blind (Subject and Rater) Controlled Study to Confirm the Effectiveness of Predictix Genetics Antidepressant -Guided Treatment in Adults With Major Depressive Disorder (MDD)
Brief Title: Confirm the Effectiveness of Predictix Genetics Antidepressant -Guided Treatment in Adults With MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taliaz Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CL-01-MCS-001
Record Dates: First submitted 2021-10-20; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Double-Blind (Subject and Rater) Controlled Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU (No Intervention): Treatment as Usual: The treating clinician will decide on what antidepressant to prescribe based on the clinical evaluation.
- PGT (Active Comparator): Predictix Guided Treatment: The treating clinician will decide on what antidepressant to prescribe based on clinical evaluation and the Predictix report
  Interventions: Device: Predictix Genetics Antidepressant

INTERVENTIONS:
Device: Predictix Genetics Antidepressant — Predictix Genetics Antidepressant (PGA) is a software tool that is intended to support a clinician in choosing the most suitable antidepressant treatment/s for an individual patient diagnosed with MDD.
  Arms: PGT

SUMMARY:
A randomized, controlled, prospective, multicenter, patient and rater blinded study with 2 arms: Treatment as Usual (TAU) and Predictix Guided Treatment (PGT). The study will compare the rate of treatment response and remission among both groups; TAU vs PGT.

DETAILED DESCRIPTION:
A randomized, controlled, prospective, multicenter, patient and rater blinded study with 2 arms: Treatment as Usual (TAU) and Predictix Guided Treatment (PGT). The study will compare the rate of treatment response and remission among both groups; TAU vs PGT.

The study will enroll up to 354 eligible patients. An interim analysis is planned after 240 evaluable subjects complete the 8-week's visit. According to the interim analysis plan, the sample size may be increased to 522.

To participate in the study the subjects must be at least 18 years old and able to give a written informed consent after an oral and written explanation of the study aims and methods. The study sample will include female and male patients with major depression diagnosis according to DSM-5 and MINI criteria. For the detailed assessment of clinical severity of specific disorder and treatment effects, the following disorder-specific rating scales will be used: Montgomery-Asberg's Depression Rating Scale (MADRS), Clinical Global Impression scale (CGI), , Patient Health Questionnaire (PHQ-9) and Patient's Global Impression (PGI). Patients will be randomized into either the Predictix Guided Treatment (PGT) group or the Treatment as Usual (TAU) group. Randomization will be stratified based on the number of previous treatment failures for the current MDD episode to ensure balance of the treatment groups. Patients will be prospectively treated with approved antidepressant medication for a period of 8 weeks (defined as a treatment cycle) during and after which they will be assessed, and treatment success or failure will be determined. Maximum desired up-titration should be reached by week 2. Concomitant treatments that are permitted include: benzodiazepines for those who had no previous hypnotic treatment - Zolpidem 10 mg at night or for anxiety -no more than 10 mg/day Diazepam or equivalent; formal psychotherapy not started within a month before the beginning of the study; non-psychopharmacologic drugs with CNS effects if the patient has been receiving a stable dose of the drug for at least one month before baseline.

Patients will be defined as responders if the decrease in MADRS scores is at least 50% compared to baseline. The remitters will be defined if the scores are less than 10 on the MADRS. Patients who do not meet these criteria will be defined as non-responders and non-remitters respectively. Following the 8 weeks, patients in the TAU group will be offered PGT in an open-label extension of the study. Patients in the TAU and PGT groups will be followed for up to an additional 2 treatment cycles (of up to 8 weeks each).

A treatment cycle will include 4 visits: Screening, Baseline (on site visit), 4 and 8 weeks (Telephone visits). At least one completed cycle per patient is required for a patient to be included in the analysis as study completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at the age of 18-75 years old at time of screening.
2. Primary diagnosis of Major Depressive Disorder (without psychosis) based on DSM-5 criteria and MINI 7.0.
3. MADRS score ≥22
4. No other causes of depressive symptoms other than MDD.
5. Ability to read, understand and sign an informed consent document.
6. Not more than 2 past failed pharmacologic interventions for the current depressive episode.
7. If subject is female and at reproductive age, she must be tested negative for pregnancy.
8. If subject is female and at reproductive age with childbearing potential (i.e., not post-menopausal or surgically sterilized) she must agree to use adequate birth control methods during the whole study duration.

Exclusion Criteria:

EXCLUSION CRITERIA

1. Patient is diagnosed with other major psychopathologies (i.e. schizophrenia, bipolar disorder, psychotic depression, geriatric depression).
2. Patient requires antipsychotic medication or mood stabilizers (other than study medication), lithium, carbamazepine, valproate and other that may have an antidepressant effect.
3. Electroconvulsive therapy (ECT) or transcranial magnetic stimulation therapy (TMS) conducted in the past or started within 90 days of screening or planned during the study.
4. Nonpsychopharmacologic drugs with CNS effects that have been taken for less than 30 days prior to baseline.
5. Subjects with a vagus nerve or deep brain stimulator.
6. Patient is at substantial suicidal risk as determined by the Mini Neuropsychiatric Interview (MINI) Suicidality subscale for suicide attempts and/or judged by the treating physician.
7. Patient has any current unstable medical condition or surgical illness.
8. Patient has history of seizure or convulsions.
9. A current status of dependence to a drug or alcohol.
10. Inadequate communication with the patient.
11. Patient has participated in another clinical study in the last 30 days preceding this study.
12. In the investigator's judgement, patient is not able to provide written informed consent and follow protocol requirements.
13. Pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 8 weeks
  Response is defined as a reduction from baseline of at least 50% (≥50%) in Montgomery-Asberg Depression Rating Scale (MADRS).

SECONDARY OUTCOMES:
Remission rate | 8 weeks
  Remission is defined as a Montgomery-Asberg Depression Rating Scale (MADRS) < 10
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) over time. | 8 weeks
  Efficacy over time
Time to response | 8 weeks
  Time to response
Clinician Global Impression (CGI) score over time | 8 weeks
  Efficacy over time

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Souery, MD, Principal Investigator — Psy Pluriel
Locations (4):
- Belgium (2):
  - Psy Pluriel, Brussels
  - Psy Pluriel, Liège
- Hospital Pitié Salpétrière, Paris, France
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taliaz D, Spinrad A, Barzilay R, Barnett-Itzhaki Z, Averbuch D, Teltsh O, Schurr R, Darki-Morag S, Lerer B. Optimizing prediction of response to antidepressant medications using machine learning and integrated genetic, clinical, and demographic data. Transl Psychiatry. 2021 Jul 8;11(1):381. doi: 10.1038/s41398-021-01488-3. PMID 34238923
- [Result] Taliaz D, Souery D. A New Characterization of Mental Health Disorders Using Digital Behavioral Data: Evidence from Major Depressive Disorder. J Clin Med. 2021 Jul 14;10(14):3109. doi: 10.3390/jcm10143109. PMID 34300275